CLINICAL TRIAL: NCT01088555
Title: Pilot Study : Effect of Sodium Thiosulfate on Urine Chemistries of Hypercalciuric Stone Formers
Brief Title: Effect of Sodium Thiosulfate on Urine Chemistries of Hypercalciuric Stone Formers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, David S. Goldfarb, M.D., PI, VA New York Harbor Healthcare System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01098
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Stones
Keywords: nephrolithiasis; calcium stones; kidney stones; hypercalciuria; sodium thiosulfate; Calcium containing kidney stones
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Hypercalciuria | interventions — sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Healthy subjects with no history of kidney stones, heart liver or kidney disease, not pregnant /lactating.
  Interventions: Drug: Sodium thiosulfate
- Stone formers (Active Comparator): History of calcium containing kidney stones, hypercalciuria on previous urine tests, no heart /liver / kidney disease, not pregnant/lactating
  Interventions: Drug: Sodium thiosulfate

INTERVENTIONS:
Drug: Sodium thiosulfate — Oral administration of sodium thiosulfate pentahydrate 5% solution (American Regent) 10ml BID x 7 days

SUMMARY:
Sodium thiosulfate may be useful to prevent recurrence of calcium-containing kidney stones. It will be studied in people with high amounts of urine calcium.

DETAILED DESCRIPTION:
The investigators study is designed as a pilot study to study the effect of STS on urine chemistries in stone formers and normal controls. It is expected to continue for a duration of 1 year and will have two groups: 20 normal controls, who are healthy subjects without known kidney disease or nephrolithiasis, and 20 subjects with documented recurrent nephrolithiasis and hypercalciuria. Patients will be recruited from Dr Goldfgarb's stone clinic at VA Hospital and controls would be voluntary participants from NYU School of Medicine. Subjects who are pregnant or nursing, taking alcohol or drugs, have known CKD or are unable to give consent would be excluded from the study. Any diuretics or citrate containing drugs would be held for a period of 2 weeks during the study period to achieve washout of the effects of those drugs on urine chemistries. Oral STS 10mmol (10ml of 25% STS) BID will be administered to both groups for 7 days; four 24 hour urine collections, 2 prior and 2 at the end of the study, would be done with all participants. A diet diary would be maintained by subjects concomitantly during the study periods. The investigators then plan to compare the two groups in terms of urine chemistries to detect any changes in these parameters with thiosulfate administration. Based on prior animal experiments and human studies with STS the investigators anticipate that it would have a favorable effect on the supersaturation of Ca oxalate/phosphate and therefore its long term use would be helpful in preventing nephrolithiasis.

ELIGIBILITY:
Inclusion Criteria:

Control arm: no longer recruiting

Hypercalciuria arm:

* Age 18-80 years old
* history of calcium-containing kidney stones
* no history of liver, heart or kidney disease (other than kidney stones)
* Non-pregnant, non-lactating
* Able to stop diuretics for a period of 1 week

Exclusion Criteria:

* Not able to sign consent
* Not satisfying any of the above criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in supersaturation of calcium oxalate / phosphate | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldfarb, MD, Principal Investigator — New York Harbor VA Medical Center
Locations (1):
- VA New York Harbor Healthcare System, New York, New York, United States